CLINICAL TRIAL: NCT06034678
Title: Evaluation of a Behavioral Intervention to Promote Food Allergy Self-Management Among Early Adolescents: The Food Allergy Mastery Program
Brief Title: Evaluation of The Food Allergy Mastery Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Northwestern University (Other); Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 30007544; R01AI168090 (NIH)
Record Dates: First submitted 2023-07-18; First posted 2023-09-13 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Food Allergy in Children
Keywords: food allergy; knowledge; management; adolescents; caregivers; social support
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food Allergy Mastery Program (Experimental): Participants randomized to the Food Allergy Mastery Program arm will participate in 6 telehealth intervention sessions with a trained mental health provider pertaining to food allergy education, food allergy management, anxiety and stress management, social situations, and self-efficacy. One of the 6 sessions is a group session with peers.
  Interventions: Behavioral: Food Allergy Mastery Program
- Usual Care (No Intervention): Participants will receive their usual allergy care.

INTERVENTIONS:
Behavioral: Food Allergy Mastery Program — Food Allergy Mastery Program sessions will be delivered by masters-level counselors as 6 45-minute biweekly telehealth or in-person sessions over a period of 3 months. Session 1 will include both youth and caregiver, Session 2 will be a group session with 5-6 youth, Session 3 will include both youth and caregiver, Sessions 4-5 will be individual youth sessions, and Session 6 will include both youth and caregiver. Sessions will incorporate a variety of formats, each based on the needs of the session content.
  Arms: Food Allergy Mastery Program

SUMMARY:
The proposed research project will evaluate a novel behavioral intervention that promotes early adolescent food allergy self-management and adjustment through 1) food allergy education, 2) problem-solving, communication, assertiveness, and anxiety management skill building, and 3) peer support.

DETAILED DESCRIPTION:
The proposed research project will evaluate a novel behavioral intervention that promotes early adolescent food allergy self-management and adjustment through 1) food allergy education, 2) problem-solving, communication, assertiveness, and anxiety management skill building, and 3) peer support. The Food Allergy Mastery (FAM) program is a 6-session food allergy self-management program that will be delivered to early adolescents with food allergy, a high-risk population that is growing in size, and a primary caregiver by a trained interventionist. The specific aims are: 1) To evaluate the intervention's impact on food allergy knowledge and self-management skills, 2) To determine the intervention's impact on food allergy self-management behavior and psychosocial functioning and healthcare utilization, and as an exploratory aim 3) to determine if early adolescents' race/ethnicity moderates response to treatment, including food allergy knowledge, skills, self-management behavior, psychosocial functioning, and healthcare utilization. The study has the potential to positively impact the health care utilization of youth with food allergy by evaluating a scalable behavioral intervention for adolescents and their caregivers. The intervention will equip youth with food allergy knowledge and self-management skills by bolstering their food allergy-related knowledge and problem-solving, social skills, and social support and attenuating food allergy anxiety. Successful development and implementation of the FAM Program that promotes the attainment of integration of food allergy into daily life has the potential to decrease health care utilization reducing emergency visits and improve food allergy-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. age 10-14 years
2. physician diagnosis (i.e., history of a reaction to the food and/or recent positive skin prick test or IgE-specific testing) of at least 1 of the 9 most common IgE-mediated food allergies (peanut, tree nut, cow's milk, egg, soy, wheat, shellfish, fish, sesame) for ≥1 year, with accompanying allergen avoidance prescribed by an allergist
3. English fluency
4. access to a device with internet access
5. either a food allergy knowledge score of <80% correct on the Food Allergy Knowledge Test (FAKT) or a food allergy impact score of ≥3 on the Food Allergy Independent Measure (FAIM).

Exclusion Criteria:

1. diagnosis of a non-IgE-mediated food allergy or food intolerance, a non-atopic chronic illness or pervasive developmental disorder/cognitive limitation
2. Current participation in psychotherapy with a therapist with food allergy expertise

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Food Allergy Knowledge | Change in Food Allergy Knowledge from Baseline to 6 Month Follow Up
  Early adolescents and caregivers will complete the Food Allergy Knowledge Test (FAKT), a -item measure of food allergy knowledge, including general clinical food allergy knowledge, avoiding exposure (i.e., cross-contact, reading labels), epinephrine auto-injector use, and signs, symptoms, and treatment of anaphylaxis. Items are scored as correct/incorrect, and a sum score is generated. Higher scores indicate greater food allergy knowledge. The FAKT was found to be highly reliable with validity analyses revealing positive score correlations with parent age, education, insurance status, access to food allergy information, and epinephrine auto-injector use.
Food Allergy Knowledge | Change in Food Allergy Knowledge from Baseline to 12 Month Follow Up
  Early adolescents and caregivers will complete the Food Allergy Knowledge Test (FAKT), a -item measure of food allergy knowledge, including general clinical food allergy knowledge, avoiding exposure (i.e., cross-contact, reading labels), epinephrine auto-injector use, and signs, symptoms, and treatment of anaphylaxis. Items are scored as correct/incorrect, and a sum score is generated. Higher scores indicate greater food allergy knowledge. The FAKT was found to be highly reliable with validity analyses revealing positive score correlations with parent age, education, insurance status, access to food allergy information, and epinephrine auto-injector use.
Food Allergy Knowledge | Change in Food Allergy Knowledge from Baseline to 18 Month Follow Up
  Early adolescents and caregivers will complete the Food Allergy Knowledge Test (FAKT), a -item measure of food allergy knowledge, including general clinical food allergy knowledge, avoiding exposure (i.e., cross-contact, reading labels), epinephrine auto-injector use, and signs, symptoms, and treatment of anaphylaxis. Items are scored as correct/incorrect, and a sum score is generated. Higher scores indicate greater food allergy knowledge. The FAKT was found to be highly reliable with validity analyses revealing positive score correlations with parent age, education, insurance status, access to food allergy information, and epinephrine auto-injector use.
Food Allergy Management Skills- Label Reading | Change in Food Allergy Management Skills- Label Reading from Baseline to 6 Month Follow Up
  Early adolescents' and caregivers' food allergy management skills will be independently assessed via direct observation of their ability to correctly read food labels and use an epinephrine auto-injector trainer. Participants will be asked to review 5 food labels for safety for themselves/their child, of which 3 food labels will not be safe and 2 food labels will be safe. A percentage correct score based on the number of labels that they correctly identify as containing or not containing allergen(s) will be calculated.
Food Allergy Management Skills- Label Reading | Change in Food Allergy Management Skills- Label Reading from Baseline to 12 Month Follow Up
  Early adolescents' and caregivers' food allergy management skills will be independently assessed via direct observation of their ability to correctly read food labels and use an epinephrine auto-injector trainer. Participants will be asked to review 5 food labels for safety for themselves/their child, of which 3 food labels will not be safe and 2 food labels will be safe. A percentage correct score based on the number of labels that they correctly identify as containing or not containing allergen(s) will be calculated.
Food Allergy Management Skills- Label Reading | Change in Food Allergy Management Skills- Label Reading from Baseline to 18 Month Follow Up
  Early adolescents' and caregivers' food allergy management skills will be independently assessed via direct observation of their ability to correctly read food labels and use an epinephrine auto-injector trainer. Participants will be asked to review 5 food labels for safety for themselves/their child, of which 3 food labels will not be safe and 2 food labels will be safe. A percentage correct score based on the number of labels that they correctly identify as containing or not containing allergen(s) will be calculated.
Food Allergy Management Skills- Epinephrine Auto-Injector Use | Change in Food Allergy Management Skills- Epinephrine Auto-Injector Use from Baseline to 6 Month Follow Up
  Participants will be asked to demonstrate how to use the epinephrine auto-injector trainer for which they have a prescription (i.e., EpiPen, AuviQ, or generic). Participants will receive a point for each of the following: removing the cap, holding it correctly, positioning it correctly on the outer thigh, "injecting" it properly, and then holding it against the thigh for the appropriate amount of time. A percentage correct score will be calculated.
Food Allergy Management Skills- Epinephrine Auto-Injector Use | Change in Food Allergy Management Skills- Epinephrine Auto-Injector Use from Baseline to 12 Month Follow Up
  Participants will be asked to demonstrate how to use the epinephrine auto-injector trainer for which they have a prescription (i.e., EpiPen, AuviQ, or generic). Participants will receive a point for each of the following: removing the cap, holding it correctly, positioning it correctly on the outer thigh, "injecting" it properly, and then holding it against the thigh for the appropriate amount of time. A percentage correct score will be calculated.
Food Allergy Management Skills- Epinephrine Auto-Injector Use | Change in Food Allergy Management Skills- Epinephrine Auto-Injector Use from Baseline to 18 Month Follow Up
  Participants will be asked to demonstrate how to use the epinephrine auto-injector trainer for which they have a prescription (i.e., EpiPen, AuviQ, or generic). Participants will receive a point for each of the following: removing the cap, holding it correctly, positioning it correctly on the outer thigh, "injecting" it properly, and then holding it against the thigh for the appropriate amount of time. A percentage correct score will be calculated.
Food Allergy Management Behaviors | Change in Food Allergy Management Behaviors from Baseline to 6 Month Follow Up
  Early adolescents will complete the Food Allergy Management 24-Hour Recall (FAM-24), a 24-hour recall interview facilitated by a research team member that asks a series of questions about each food they ate during the previous day. Participants report on the time of the meal/snack, where they ate (e.g., school, home, a restaurant), whether an adult was present, whether epinephrine was available, and if so, where it was located (e.g., on person, in another room). They also report if they had an allergic reaction. For each individual food eaten during the meal/snack, participants report what the food was, whether they ate it before, whether it was verified as allergen-free, how it was verified (e.g., prepared at home, read the label, asked about ingredients), and who verified it (e.g., child, parent, teacher, another adult). Participants can endorse multiple methods of allergen-free verification and multiple people who completed the verification.
Food Allergy Management Behaviors | Change in Food Allergy Management Behaviors from Baseline to 12 Month Follow Up
  Early adolescents will complete the Food Allergy Management 24-Hour Recall (FAM-24), a 24-hour recall interview facilitated by a research team member that asks a series of questions about each food they ate during the previous day. Participants report on the time of the meal/snack, where they ate (e.g., school, home, a restaurant), whether an adult was present, whether epinephrine was available, and if so, where it was located (e.g., on person, in another room). They also report if they had an allergic reaction. For each individual food eaten during the meal/snack, participants report what the food was, whether they ate it before, whether it was verified as allergen-free, how it was verified (e.g., prepared at home, read the label, asked about ingredients), and who verified it (e.g., child, parent, teacher, another adult). Participants can endorse multiple methods of allergen-free verification and multiple people who completed the verification.
Food Allergy Management Behaviors | Change in Food Allergy Management Behaviors from Baseline to 18 Month Follow Up
  Early adolescents will complete the Food Allergy Management 24-Hour Recall (FAM-24), a 24-hour recall interview facilitated by a research team member that asks a series of questions about each food they ate during the previous day. Participants report on the time of the meal/snack, where they ate (e.g., school, home, a restaurant), whether an adult was present, whether epinephrine was available, and if so, where it was located (e.g., on person, in another room). They also report if they had an allergic reaction. For each individual food eaten during the meal/snack, participants report what the food was, whether they ate it before, whether it was verified as allergen-free, how it was verified (e.g., prepared at home, read the label, asked about ingredients), and who verified it (e.g., child, parent, teacher, another adult). Participants can endorse multiple methods of allergen-free verification and multiple people who completed the verification.
Food Allergy Quality of Life- Child Self Report | Change in Food Allergy Quality of Life- Child Self Report from Baseline to 6 Month Follow Up
  Early adolescents will complete the Food Allergy Quality of Life Questionnaire - Child Form (8-12 years) (FAQLQ-CF), a validated 10-item measure, or the Food Allergy Quality of Life Questionnaire - Teenager Form (13-17 years) (FAQLQ-TF), a validated 10-item measure. Participants only complete the questionnaire appropriate for their age. Items for these scales are rated on a 7-point Likert scale; subscale and total scores are generated with higher scores indicating greater food allergy anxiety and impact of food allergy on quality of life. Score range is 0-60.
Food Allergy Quality of Life- Child Self-Report | Change in Food Allergy Quality of Life- Child Self Report from Baseline to 12 Month Follow Up
  Early adolescents will complete the Food Allergy Quality of Life Questionnaire - Child Form (8-12 years) (FAQLQ-CF), a validated 10-item measure, or the Food Allergy Quality of Life Questionnaire - Teenager Form (13-17 years) (FAQLQ-TF), a validated 10-item measure. Participants only complete the questionnaire appropriate for their age. Items for these scales are rated on a 7-point Likert scale; subscale and total scores are generated with higher scores indicating greater food allergy anxiety and impact of food allergy on quality of life. Score range is 0-60.
Food Allergy Quality of Life- Child Self-Report | Change in Food Allergy Quality of Life- Child Self Report from Baseline to 18 Month Follow Up
  Early adolescents will complete the Food Allergy Quality of Life Questionnaire - Child Form (8-12 years) (FAQLQ-CF), a validated 10-item measure, or the Food Allergy Quality of Life Questionnaire - Teenager Form (13-17 years) (FAQLQ-TF), a validated 10-item measure. Participants only complete the questionnaire appropriate for their age. Items for these scales are rated on a 7-point Likert scale; subscale and total scores are generated with higher scores indicating greater food allergy anxiety and impact of food allergy on quality of life. Score range is 0-60.
Food Allergy Quality of Life- Parent Proxy | Change in Food Allergy Quality of Life- Parent Proxy from Baseline to 6 Month Follow Up
  Caregivers will complete the Food Allergy Quality of Life Questionnaire - Parent Form (FAQLQ-PF), a validated 10-item measure of parents' perceptions of their child's quality of life. Items for these scales are rated on a 7-point Likert scale; subscale and total scores are generated with higher scores indicating greater food allergy anxiety and impact of food allergy on quality of life. Score range is 0-60.
Food Allergy Quality of Life- Parent Proxy | Change in Food Allergy Quality of Life- Parent Proxy from Baseline to 12 Month Follow Up
  Caregivers will complete the Food Allergy Quality of Life Questionnaire - Parent Form (FAQLQ-PF), a validated 10-item measure of parents' perceptions of their child's quality of life. Items for these scales are rated on a 7-point Likert scale; subscale and total scores are generated with higher scores indicating greater food allergy anxiety and impact of food allergy on quality of life. Score range is 0-60.
Food Allergy Quality of Life- Parent Proxy | Change in Food Allergy Quality of Life- Parent Proxy from Baseline to 18 Month Follow Up
  Caregivers will complete the Food Allergy Quality of Life Questionnaire - Parent Form (FAQLQ-PF), a validated 10-item measure of parents' perceptions of their child's quality of life. Items for these scales are rated on a 7-point Likert scale; subscale and total scores are generated with higher scores indicating greater food allergy anxiety and impact of food allergy on quality of life. Score range is 0-60.
Food Allergy Impact | Change in Food Allergy Impact from Baseline to 6 Month Follow Up
  Children will complete the Food Allergy Independent Measure (FAIM), a 6-item measure of children's perceptions of risk of allergen exposure, chance of a severe reaction, chance of dying, and ability to engage in proper treatment, which generates a total score. Scores can range from 0-6; higher scores indicate more impact of food allergy on daily life.
Food Allergy Impact | Change in Food Allergy Impact from Baseline to 12 Month Follow Up
  Children will complete the Food Allergy Independent Measure (FAIM), a 6-item measure of children's perceptions of risk of allergen exposure, chance of a severe reaction, chance of dying, and ability to engage in proper treatment, which generates a total score. Scores can range from 0-6; higher scores indicate more impact of food allergy on daily life.
Food Allergy Impact | Change in Food Allergy Impact from Baseline to 18 Month Follow Up
  Children will complete the Food Allergy Independent Measure (FAIM), a 6-item measure of children's perceptions of risk of allergen exposure, chance of a severe reaction, chance of dying, and ability to engage in proper treatment, which generates a total score. Scores can range from 0-6; higher scores indicate more impact of food allergy on daily life.
Frequency of Treatment for Allergic Reactions | Change in Frequency of Treatment for Allergic Reactions from Baseline to 6 Month Follow Up
  Participants will report on the frequency of treatment for allergic reactions in the past 6 months. This information will also be assessed by study staff via clinic chart review.
Frequency of Treatment for Allergic Reactions | Change in Frequency of Treatment for Allergic Reactions from Baseline to 12 Month Follow Up
  Participants will report on the frequency of treatment for allergic reactions in the past 6 months. This information will also be assessed by study staff via clinic chart review.
Frequency of Treatment for Allergic Reactions | Change in Frequency of Treatment for Allergic Reactions from Baseline to 18 Month Follow Up
  Participants will report on the frequency of treatment for allergic reactions in the past 6 months. This information will also be assessed by study staff via clinic chart review.
Frequency of Allergy Appointments | Change in Frequency of Allergy Appointments from Baseline to 6 Month Follow Up
  Participants will report on the frequency of allergy appointments in the past 6 months. This information will also be assessed by study staff via clinic chart review.
Frequency of Allergy Appointments | Change in Frequency of Allergy Appointments from Baseline to 12 Month Follow Up
  Participants will report on the frequency of allergy appointments in the past 6 months. This information will also be assessed by study staff via clinic chart review.
Frequency of Emergency Room/Urgent Care Visits for Allergic Reactions | Change in Frequency of Emergency Room/Urgent Care Visits for Allergy Reactions from Baseline to 6 Month Follow Up
  Participants will report on the frequency of emergency room/urgent care visits for allergic reactions in the past 6 months. This information will also be assessed by study staff via clinic chart review.
Frequency of Allergy Appointments | Change in Frequency of Allergy Appointments from Baseline to 18 Month Follow Up
  Participants will report on the frequency of allergy appointments in the past 6 months. This information will also be assessed by study staff via clinic chart review.
Frequency of Emergency Room/Urgent Care Visits for Allergic Reactions | Change in Frequency of Emergency Room/Urgent Care Visits for Allergy Reactions from Baseline to 12 Month Follow Up
  Participants will report on the frequency of emergency room/urgent care visits for allergic reactions in the past 6 months. This information will also be assessed by study staff via clinic chart review.
Frequency of Emergency Room/Urgent Care Visits for Allergic Reactions | Change in Frequency of Emergency Room/Urgent Care Visits for Allergy Reactions from Baseline to 18 Month Follow Up
  Participants will report on the frequency of emergency room/urgent care visits for allergic reactions in the past 6 months. This information will also be assessed by study staff via clinic chart review.

SECONDARY OUTCOMES:
Social Support | Change in Social Support from Baseline to 6 Month Follow Up
  Early adolescents will complete the Multidimensional Scale of Perceived Social Support (MSPSS) to measure agreement with statements of general subjectively assessed social support from friends, family, and a significant other. The MSPSS consists of 12 items that assess perceived social support. Respondents elect responses on a Likert-type scale from 0 ("Very Strongly Disagree") to 6 ("Very Strongly Agree"). Total scores are computed by calculating the mean of all items, and higher scores indicate greater perceived social support. Score range is 0-6.
Social Support | Change in Social Support from Baseline to 12 Month Follow Up
  Early adolescents will complete the Multidimensional Scale of Perceived Social Support (MSPSS) to measure agreement with statements of general subjectively assessed social support from friends, family, and a significant other. The MSPSS consists of 12 items that assess perceived social support. Respondents elect responses on a Likert-type scale from 0 ("Very Strongly Disagree") to 6 ("Very Strongly Agree"). Total scores are computed by calculating the mean of all items, and higher scores indicate greater perceived social support. Score range is 0-6.
Social Support | Change in Social Support from Baseline to 18 Month Follow Up
  Early adolescents will complete the Multidimensional Scale of Perceived Social Support (MSPSS) to measure agreement with statements of general subjectively assessed social support from friends, family, and a significant other. The MSPSS consists of 12 items that assess perceived social support. Respondents elect responses on a Likert-type scale from 0 ("Very Strongly Disagree") to 6 ("Very Strongly Agree"). Total scores are computed by calculating the mean of all items, and higher scores indicate greater perceived social support. Score range is 0-6.
Food Allergy Self-Efficacy | Change in Food Allergy Self-Efficacy from Baseline to 6 Month Follow Up
  Early adolescents and caregivers will each complete the Food Allergy Self-Efficacy Scale (FASE), a 21-item measure that uses a 100-point visual analog scale. Higher scores indicate a greater degree of confidence in one's ability to manage food allergies. Score range is 0-100. The FASE is valid and reliable among parents.
Food Allergy Self-Efficacy | Change in Food Allergy Self-Efficacy from Baseline to 12 Month Follow Up
  Early adolescents and caregivers will each complete the Food Allergy Self-Efficacy Scale (FASE), a 21-item measure that uses a 100-point visual analog scale. Higher scores indicate a greater degree of confidence in one's ability to manage food allergies. Score range is 0-100. The FASE is valid and reliable among parents.
Food Allergy Self-Efficacy | Change in Food Allergy Self-Efficacy from Baseline to 18 Month Follow Up
  Early adolescents and caregivers will each complete the Food Allergy Self-Efficacy Scale (FASE), a 21-item measure that uses a 100-point visual analog scale. Higher scores indicate a greater degree of confidence in one's ability to manage food allergies. Score range is 0-100. The FASE is valid and reliable among parents.
Food Allergy Anxiety | Change in Food Allergy Anxiety from Baseline to 6 Month Follow Up
  Early adolescents and caregivers will each complete the Scale of Food Allergy Anxiety (SOFAA), a 21-item measure that uses a Likert scale (0=Never to 4=Almost Always). Higher scores indicate more food allergy anxiety. Score range is 0-84. The SOFAA is valid and reliable among parents.
Food Allergy Anxiety | Change in Food Allergy Anxiety from Baseline to 12 Month Follow Up
  Early adolescents and caregivers will each complete the Scale of Food Allergy Anxiety (SOFAA), a 21-item measure that uses a Likert scale (0=Never to 4=Almost Always). Higher scores indicate more food allergy anxiety. Score range is 0-84. The SOFAA is valid and reliable among parents.
Food Allergy Anxiety | Change in Food Allergy Anxiety from Baseline to 18 Month Follow Up
  Early adolescents and caregivers will each complete the Scale of Food Allergy Anxiety (SOFAA), a 21-item measure that uses a Likert scale (0=Never to 4=Almost Always). Higher scores indicate more food allergy anxiety. Score range is 0-84. The SOFAA is valid and reliable among parents.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Herbert, PhD, Principal Investigator — Childrens National Hospital
Locations (1):
- Childrens' National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No